CLINICAL TRIAL: NCT02727712
Title: Studies of Application of Combined General Anesthesia and Bilateral Thoracic Paravertebral Block by Ropivacaine in Patients Undergoing Off-pump Coronary Artery Bridge Graft - a Random Double Blind Controlled Study
Brief Title: Studies of Application of Combined General Anesthesia and Bilateral TPVB in OPCABG
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20160131
Record Dates: First submitted 2016-02-22; First posted 2016-04-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Coronary Heart Disease
Keywords: coronary artery bypass graft; thoracic paravertebral block
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TPVB T2/3+T5/6+GA (Experimental): the group A of patients has been received bilateral thoracic paravertebral block (TPVB T2/3+T5/6) by ropivacaine(0.3%,10ml*4), before general anesthesia management
  Interventions: Procedure: bilateral thoracic paravertebral block; Device: Transesophageal Echocardiography（TEE）; Device: Lung protection measure during the surgery（Dräger Primus）; Drug: Anesthesia drugs during the surgery
- TPVB T3/4+GA (Experimental): the group Bof patients has been received bilateral thoracic paravertebral block (TPVB 3/4) by ropivacaine(0.3%,10ml*4), before general anesthesia management Device: The use of Transesophageal Echocardiography（TEE）、STAT PROFILE® and Haemonetics® during the surgery
  Interventions: Device: Transesophageal Echocardiography（TEE）; Device: Lung protection measure during the surgery（Dräger Primus）; Drug: Anesthesia drugs during the surgery; Procedure: thoracic paravertebral block
- GA (Placebo Comparator): group C under control (without TPVB)program Device: The use of Transesophageal Echocardiography（TEE）、STAT PROFILE® and Haemonetics® during the surgery
  Interventions: Device: Transesophageal Echocardiography（TEE）; Device: Lung protection measure during the surgery（Dräger Primus）; Drug: Anesthesia drugs during the surgery

INTERVENTIONS:
Procedure: bilateral thoracic paravertebral block — group A under TPVB((TPVB T2/3+T5/6) by ropivacaine(0.3%,10ml*4)program
  Arms: TPVB T2/3+T5/6+GA
Device: Transesophageal Echocardiography（TEE） — 1. Apply Transesophageal Echocardiography（TEE）after anesthesia induction and draw 400ml autologous blood (Haemonetics®)used for the postoperative transfusion;
  2. Goal-directed fluid management
Device: Lung protection measure during the surgery（Dräger Primus） — Protective ventilation strategy(Low tidal volume about 6~7ml/kg, joint use of PEEP)
Drug: Anesthesia drugs during the surgery — 1. Bilateral thoracic paravertebral block before induction of anesthesia;
  2. Fast channel anesthesia • Induction use Sufentanil 0.5~1ug/kg, Vecuronium for Injection 0.15mg/kg and Etomidate 0.2~0.6mg/kg; ②. Maintain use Sufentanil Hydrochloride for Injection 0.01~0.04ug/kg•min, Sevoflurane 0.5~1.5MAC（minimum alveolar concentration） and Infusing Dexmedetomidine which load dose 0.5μg/kg in 10min then changed into 0.5-1.0μg/kg•h,Vecuronium 0.06~0.12mg/kg•h; ③. Intravenous hydromorphone Hydrochloride Injection 0.15mg/kg before surgery over.
Procedure: thoracic paravertebral block — group B under(TPVB T3/4)by ropivacaine(0.3%,20ml*2)program
  Arms: TPVB T3/4+GA

SUMMARY:
This study intends to compare the combination of general anesthesia (GA) and single-shot bilateral thoracic paravertebral block (TPVB) by ropivacaine in the patients undergoing off-pump coronary artery bypass surgery ( OPCAB) with traditional general anesthesia (GA) perioperative management of patients, committed to reducing patient's physical and psychological stress by surgical trauma, achieve the purpose of fast recovery, in order to establish an more effective perioperative management during off-pump coronary artery bypass surgery, improve patients' satisfaction and to accelerate postoperative rehabilitation safely.

DETAILED DESCRIPTION:
This study intends to compare the combination of general anesthesia (GA) and single-shot bilateral thoracic paravertebral block (TPVB) by ropivacaine in the patients undergoing off-pump coronary artery bypass surgery ( OPCAB) with traditional general anesthesia (GA) perioperative management of patients, committed to reducing patient's physical and psychological stress by surgical trauma, achieve the purpose of fast recovery, in order to establish an more effective perioperative management during off-pump coronary artery bypass surgery, improve patients' satisfaction and to accelerate postoperative rehabilitation safely. Patients included in the study (approximately 60 cases) will be randomly divided into PVB(T2/3+T5/6)+GA experimental group (A), PVB(T3/4)+GA experimental group (B)the conventional GA control group (C). All groups received the preoperative preparation, anesthesia and postoperative treatment according to the traditional manner, the group A of patients has been received bilateral thoracic paravertebral block (TPVB T2/3+T5/6) by ropivacaine(0.3%,10ml*4), group B will received bilateral thoracic paravertebral block (TPVB T3/4)by ropivacaine(0.3%,20ml*2).,while the group C will received the conventional general anesthesia management without block.

ELIGIBILITY:
Inclusion Criteria:

* Heart function grade II - III (Using the cardiac function classification method formulated by American Heart Disease Institute)
* The in - hospital was treated with off pump coronary artery bypass grafting（CABG) operation and general anesthesia.
* Had a good cognition, and signed the informed consent.
* Aged between 35 and 80.
* The age, clinical examination and other generally situation of the two groups of patients had no statistical significance.

no merger of valvular disease left ventricular ejection fraction > 40%, do not need intraaortic balloon counterpulsation support, without spinal deformity, no vertebral side clearance space-occupying lesions

Exclusion Criteria:

* Combined with other blood coagulation dysfunction, serious brain, liver and kidney dysfunction, endocrine system diseases and serious infectious disease.
* Patients with severe mental disorders cannot cooperate with the treatment.
* Emergency operation
* Have taboo of Echocardiography and pulmonary catheterization by echocardiography.
* Allergic to Local anesthetics drug.
* Suspected or had alcohol, drug abuse history.
* Spinal or paravertebral lesions.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Fasting blood glucose | baseline and 4 days
  1day before and 4days after operation
Blood Lactic Acid | baseline and 4 days
  1day before and 4days after operation
Creatine kinase isoenzymes | baseline and 4 days
  1day before and 4days after operation
Myoglobin | baseline and 4 days
  1day before and 4days after operation
Troponin I | baseline and 4 days
  1day before and 4days after operation
White Blood Cell | baseline and 4 days
  1day before and 4days after operation
C-reactive protein | baseline and 4 days
  1day before and 4days after operation
N-terminal B-type natriuretic peptide（NT-proBNP) | baseline and 4 days
  1day before and 4days after operation

SECONDARY OUTCOMES:
Perioperative major adverse events | From pre-surgery to discharge, up to 4 weeks
Perioperative use of vasoactive drug species | From pre-surgery to discharge, up to 4 weeks
Vasoactive drugs Support Hours | From the start of drugs to stop them, up to 4 weeks
Time after deactivation of vasoactive drugs | From the end of surgery to the deactivation of vasoactive drugs, up to 4 weeks
Postoperative tracheal tube time | From the end of surgery to the removal of tracheal tube, up to 4 weeks
Duration of mechanical ventilation after surgery | From the end of surgery to the recovery of spontaneous breathing, up to 4 weeks
The time after the ICU until discharge | From leaving the ICU to discharge from hospital, up to 4 weeks
Length of ICU stay | From ICU admission to discharge from ICU, up to 4 weeks
Recovery time | From the end of surgery to recover, up to 4 weeks
Time to first bowel movement | From the end of surgery to first bowel movement, up to 2 weeks
Postoperative to normal eating time | From the end of surgery to normal eating, up to 2 weeks
The total length of hospital stay | From admission to discharge, up to 5 weeks
Visual analog pain score | From the end of surgery, up to 48 hours
Ramsay score | From the end of surgery, up to 48 hours

OTHER OUTCOMES:
The scores of mini-mental state examination | From the end of surgery, up to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: e wang, phD, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Olivier JF, Bracco D, Nguyen P, Le N, Noiseux N, Hemmerling T; Perioperative Cardiac Surgery Research Group (PeriCARG). A novel approach for pain management in cardiac surgery via median sternotomy: bilateral single-shot paravertebral blocks. Heart Surg Forum. 2007;10(5):E357-62. doi: 10.1532/HSF98.20071082. PMID 17855198
- [Result] Ganapathy S, Murkin JM, Boyd DW, Dobkowski W, Morgan J. Continuous percutaneous paravertebral block for minimally invasive cardiac surgery. J Cardiothorac Vasc Anesth. 1999 Oct;13(5):594-6. doi: 10.1016/s1053-0770(99)90015-0. No abstract available. PMID 10527232
- [Result] Mehta Y, Arora D, Sharma KK, Mishra Y, Wasir H, Trehan N. Comparison of continuous thoracic epidural and paravertebral block for postoperative analgesia after robotic-assisted coronary artery bypass surgery. Ann Card Anaesth. 2008 Jul-Dec;11(2):91-6. doi: 10.4103/0971-9784.41576. PMID 18603748
- [Result] Dhole S, Mehta Y, Saxena H, Juneja R, Trehan N. Comparison of continuous thoracic epidural and paravertebral blocks for postoperative analgesia after minimally invasive direct coronary artery bypass surgery. J Cardiothorac Vasc Anesth. 2001 Jun;15(3):288-92. doi: 10.1053/jcan.2001.23271. PMID 11426357